CLINICAL TRIAL: NCT05889000
Title: Quality of Life Questionnaire and Disease Severity Scale for Patients With Chronic Pelvic Venous Disorders: Design and Validation
Brief Title: Quality of Life Questionnaire and Disease Severity Scale
Status: Completed | Type: Observational
Sponsor: Kazan State Medical University (Other)
Collaborators: Interregional Clinical Diagnostic Center, Russia (Other)
Responsible Party: Principal Investigator, Rustem V. Akhmetzyanov, MD, PhD., Associate Professor of the Department of Cardiovascular and Endovascular Surgery, Kazan State Medical University
Other Study IDs: 10012022
Record Dates: First submitted 2023-05-24; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Pelvic Congestion Syndrome
Keywords: quality of life questionnaire; chronic pelvic venous disorders; Pelvic Varicose Veins Questionnaire; pelvic congestion syndrome; validation; Pelvi Venous Clinical Severity Score
MeSH Terms: interventions — Coping Responses Inventory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- main group: 304 patients with verified CPVD
  Interventions: Other: questionnaire responses
- comparison group: 93 participants without signs of CPVD.
  Interventions: Other: questionnaire responses

INTERVENTIONS:
Other: questionnaire responses — questionnaire responses - Pelvic Varicose Veins Questionnaire (PVVQ) and Pelvic Venous Clinical Severity Score (PVCSS)

SUMMARY:
There are currently no specific validated patient-centric tools for the clinical evaluation of patients with chronic pelvic venous disorders (CPVD). The study involves the development and validation of a questionnaire for the quality of life and a scale of disease severity for a patient with pelvic venous disease.

DETAILED DESCRIPTION:
This retrospective study will include patients with pelvic varicose veins seen between 2018 and 2020.

2 groups of patients will be formed. The main group will be women with verified CPVD, the comparison group - 93 participants without signs of CPVD.

All patients will respond to the previously developed Pelvic Varicose Veins Questionnaire (PVVQ) and Pelvic Venous Clinical Severity Score (PVCSS) as submitted questionnaires.

Validation of the PVVQ questionnaire and the PVCSS scale will be carried out in accordance with the methodology for studying the quality of life and clinical scales in accordance with international standards. The main psychometric properties of both instruments in terms of validity, reliability and sensitivity will be assessed.

The validation protocol will include certain steps: 1) pre-testing, 2) assessing the reliability of the questionnaire, 3) assessing the validity, 4) assessing the sensitivity.

1. Preliminary testing. For preliminary testing, patients will fill out questionnaires, followed by finding out how clear the questions asked are, how accurate and ethical the formulations are, in their opinion. The convenience of working with the questionnaire from the point of view of the research doctor will also be assessed.
2. Reliability assessment. The reliability assessment will be carried out according to three criteria - internal consistency, discriminant validity and internal consistency.

   To assess the degree of internal consistency, the Cronbach's alpha coefficient will be used, which is calculated by the formula: α = N * r / (1 + r * (N - 1)), where N is the number of components under study, r is the average correlation coefficient between the components. The study will assess the reliability of the questionnaire and the scale as a whole, as well as the impact on the overall reliability of each individual domain. Domain correlation will be assessed using Spearman's rank correlation method (r).

   To assess discriminant validity, the level of quality of life and disease severity of patients with VBT will be compared with similar levels of healthy participants.

   Assessment of internal consistency will be performed by retesting stable patients without treatment after 14 days, followed by calculation of Cronbach's alpha.
3. Assessment of validity. To assess the validity, the reliability of the construct will be studied by determining the criterion validity, i.e. identifying the correlation coefficient or relationships between the scales of both questionnaires with some external criterion. The scales of the SF-36 questionnaire will be used as external criteria for assessing the quality of life, and elements of visual analogue scales will be used to assess the severity of the disease.

   To study the degree of representation of the studied psychological construct in the test results, both types of construct validity will be determined: convergent and discriminant.
4. Sensitivity assessment. To assess the sensitivity, a comparison of the indicators of the questionnaire questionnaires at the points before treatment and 2 months after the treatment will be carried out.

Based on this examination of the data, objective information on the validity, reliability and sensitivity of PVVQ and PVCSS will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* presence of PVV;
* completed Patient Informed Consent Form;
* age from 18 to 70 years;
* ability to understand and answer the questions of the proposed questionnaire.

Exclusion Criteria:

* absence of confirmed PVV;
* lack of Patient Informed Consent Form;
* under the age of 18 or over 70 years old;
* pregnancy at any stage and 12-month postpartum period;
* presence of a gynecological or other concomitant (urological, neurological, procto-logical, etc.) significant pathology that has similar clinical symptoms with CPVD and re-quires specific treatment;
* presence of severe concomitant gastrointestinal or hematopoietic system pathology, terminal stages of cardiovascular, respiratory, renal and hepatic failure, stage IV malignant tumor, obliterating diseases of lower limbs arteries;
* dementia and other mental disorders that limit the ability to understand the essence of the research, fill out Patient Informed Consent Form and answer the questionnaire

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients attending primary care
Sampling Method: Probability Sample
Enrollment: 397 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
internal consistency assessment | At baseline
  To assess the degree of internal consistency, the Cronbach's alpha coefficient will be used, which is calculated by the formula: α = N * r / (1 + r * (N - 1)), where N is the number of components under study, r is the average correlation coefficient between the components. The study will assess the reliability of the questionnaire and the scale as a whole, as well as the impact on the overall reliability of each individual domain. Domain correlation will be assessed using Spearman's rank correlation method (r).
discriminant validity evaluation internal consistency score | At baseline
  To assess discriminant validity, the level of quality of life and disease severity of patients with CPVD will be compared with similar levels of healthy participants.
internal consistency score | At baseline and after 14 days
  Assessment of internal consistency will be performed by retesting stable patients without treatment after 14 days, followed by calculation of Cronbach's alpha.
determination of criterion validity | At baseline
  To assess the validity, the reliability of the construct will be studied by determining the criterion validity, i.e. identifying the correlation coefficient or relationships between the scales of both questionnaires with some external criterion. The scales of the SF-36 questionnaire will be used as external criteria for assessing the quality of life, and elements of visual analogue scales will be used to assess the severity of the disease.
Sensitivity assessment. | At baseline and after 2 months
  To assess the sensitivity, a comparison of the indicators of the questionnaire questionnaires at the points before treatment and 2 months after the treatment will be carried out.

CONTACTS AND LOCATIONS:
Overall Officials: Aigul A Mutygullina, PhD, Study Director — Kazan State Medical University
Locations (1):
- State Medical University, Kazan', Tatarstan Republic, Russia